CLINICAL TRIAL: NCT03332719
Title: Multicentric Evaluator-blinded Randomized Non-inferiority Study, to Asses the Compared Efficacy, Safety and Immunogenicity of Enerceptan® With Enbrel® in Combination With Methotrexate for the Treatment of Patients With Rheumatoid Arthritis
Brief Title: Efficacy, Safety and Immunogenicity of Enerceptan Compared to Enbrel in Rheumatoid Arthritis
Acronym: GEMENE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gema Biotech S.A. (Industry)
Collaborators: QUID Quality in Drugs and Devices Latin American Consulting SRL (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GEMENE001
Record Dates: First submitted 2016-04-21; First posted 2017-11-06 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Etanercept; Methotrexate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Enbrel® (Active Comparator): Enbrel® 50 mg injectable solution in autoinjector SureClick® contains: 50 mg etanercept and excipients/Once a week Methotrexate 15 to 25 mg /Once a week
  Interventions: Biological: Etanercept; Drug: Methotrexate
- Enerceptan®. (Experimental): Enerceptan®. Injectable Solution in prefilled syringes Source: GEMABIOTECH S. A. Formulation per unit: 1,0 ml of Enerceptan® contains 50 mg solution of Etanercept /Once a week Methotrexate 15 to 25 mg /Once a week
  Interventions: Biological: Etanercept; Drug: Methotrexate

INTERVENTIONS:
Biological: Etanercept
Drug: Methotrexate

SUMMARY:
The purpose of this study is to asses the compared efficacy, safety and immunogenicity of ENERCEPTAN® with ENBREL® in combination with Methotrexate for the treatment of patients with rheumatoid arthritis.

DETAILED DESCRIPTION:
Randomized, , non-inferiority, two parallel arms, 32 weeks, blind for the assessor.

Subjects should be with inadequate response to methotrexate with stable dosis ≥ 15 and ≤ 25 mg/week 28 days before randomization.

Randomization will be 2:1 Enerceptan® to Enbrel® with concomitant medication of MTX

ELIGIBILITY:
Inclusion Criteria:

1. Adult men and women over 18 years, who present moderate to severe active RA (rheumatoid arthritis) , diagnosed according to ACR/ EULAR 2010 criteria, who have failed prior MTX (methotrexate) therapy. Functional class I to III.
2. Moderate to severe disease activity, according to DAS28 (erythrosedimentation) ≥ 3.2.
3. Must have at least a minimum of 6 tender joints and 8 swollen joints. If a patient has a joint surgery prior to the study, this joint is considered not evaluable throughout the study development.
4. Must have at least, one erosion in the baseline radiograph. Local assessment centers either radiologist or rheumatologist to decide on this criterion will be accepted.
5. Medical Indication to incorporate a biological treatment in their therapy.
6. Treatment with MTX for at least 3 months on dose ≥15 mg/ week, stable over the last 28 days before the Day 1. Doses lower than 15 mg and greater or equal than 10 mg/ week are accepted in cases with previously documented intolerance.
7. Subjects who have previously received treatment with a biologic (approved or investigational) except etanercept, may participate as long as the corresponding washout time has elapsed prior to the screening interview: At least

   1. 8 weeks for infliximab (T1/2 8 to 9.5 days) and for tocilizumab (T1/2 3to 12 days)
   2. 10 weeks for adalimumab (T1/2 10 to 20 days), Golimumab (T1/2 11 to 14 days), certolizumab (T1/2 14 days), abatacept (T1/2 14 days),
   3. 1 year for Rituximab (T1/2 77,5 days)
   4. 5 T1/2 for any other biological product, used for the treatment of rheumatoid arthritis, wether it has been used or not for research.
   5. Subjects who are receiving leflunomide must have a previous washout of 8 weeks before Day 1, except had have treatment with colestyramine, according to manufacturer indications.
   6. Can receive non steroidal anti inflammatory drugs (NSAIDs) or oral corticoids in doses < 10 mg of prednisone, but treatment must have been stable over the last 28 days.

      8 Subjects must be able to self-inject or willing to have a previously assigned caregiver do it for them.

      9 Subjects must be able to meet the schedule of visits, understand and comply with other protocol requirements.

      10 Women of childbearing age must commit to be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 12 weeks after the last dose of Enbrel®/Enerceptan®. Suitable methods of contraception are oral contraceptives, IUDs (intrauterine device) , bilateral tubal ligation, vasectomy or double barrier methods such as condoms or spermicidal diaphragm, sponge, contraceptive foam or gel, heterosexual abstinence. Men should not conceive up to 12 weeks after stopping the MTX

      11 Informed consent must be signed before making any study-specific procedure.

Exclusion Criteria:

1. Simultaneous treatment with other investigational drug or participation in another clinical study that the investigator considers inadvisable.
2. Women who are pregnant or breastfeeding.
3. Past history of nonresponsive to TNF (tumor necrosis factor) blocking agents or other biologic treatment.
4. Chronic antibiotic therapy, if the investigator considers this may affect the safety of the subject or the assessment of the study results.
5. Any previous or current serious medical conditions that, in the opinion of the investigator, constitute a contraindication for the study treatment, as:
6. Administration of vaccines:

   1. Subjects who have received a live attenuated vaccine within 3 months prior to the randomization Visit (for example, varicella-zoster, oral polio, rabies, yellow fever vaccines.)
   2. Subjects who have received the BCG (bacillus Calmette-Guerin) vaccine within 12 months before the Selection.
7. Presence of :

   a. At the time of the inclusion i. Active infections. ii. Fever (≥38 °C) or active, chronic or recurrent infections that require treatment with antibiotics, antiviral, or anti-fungal medications within 4 weeks prior to Screening Visit, or history of frequent recurrent infections unacceptable to the investigator's opinion.

   iii. Non-healing infected skin ulcers. b. In the previous time: i. Background of recurrent bacterial, viral, fungal (excluding superficial infections or nail bed mycosis), mycobacterial or other severe infections within the last month previous to selection.

   ii. Hospitalization for infection or Subjects who have received antibiotics intravenously within the last month or orally within the last 2 weeks.

   iii. Subjects with herpes zoster in the last 2 months.
8. Past history of drug or alcohol abuse within the last year prior to the Screening Visit.
9. Known hypersensitivity to the study drug or history of severe allergy or anaphylactic reaction to monoclonal antibodies or fusion or human proteins.
10. Any condition that, in the investigator opinion, would not allow compliance with the guidelines of the study by the patient.
11. The subject presents absolute contraindications for the use of etanercept, according to the prospectus
12. Presence of significant laboratory abnormalities in the screening visit.

Ages: 19 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2016-02; Primary Completion 2017-03 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
ACR (American College of Rheumatology) 20 | 32 weeks of treatment
  The percentage of patients who achieved ACR20 at Week 32 is the primary end point. Signs and symptoms are assessed with a composite rating scale of the ACR (American College of
  Rheumatology) that includes 7 variables:
  * Tender Joints Count
  * Swollen Joints Count
  * Levels of an acute phase reactant (CRP level)
  * Patient's assessment of pain
  * Patient's global assessment of disease activity
  * Physician's global assessment of disease activity
  * Patient's assessment of physical function

SECONDARY OUTCOMES:
ACR (American College of Rheumatology) 50 | 32 weeks of treatment
  ACR50 is defined as the percentage of patients who achieve at least 50% improvement in both tender joint count and swollen joint count, and at least 50% improvement in at least 3 of the 5 other assessments.
ACR (American College of Rheumatology) 70 | 32 weeks of treatment
  ACR70 is defined as the percentage of patients who achieve at least 70% improvement in both tender joint counts and swollen joint counts and at least 70% improvement in at least 3 of the 5 other assessments of the ACR
DAS (Disease activity state) | 32 weeks of treatment
  It will be measured using the DAS (Disease activity state) 28. DAS28 is a composite score that includes 4 variables:
  * Tender Joints Count (based on 28 joints)
  * Swollen Joints Count (based on 28 joints)
  * Patient's global assessment of disease activity
  * Marker of inflammation: C REACTIVE PROTEIN
EULAR (European League Against Rheumatism) response criteria | 32 weeks of treatment
  * Good response = Percentage of patients with an improvement of >1.2 and a present DAS score ≤3.2.
  * Moderate response = Percentage of patients with either an improvement of >0.6 to ≤1.2 and a present score ≤5.1, or an improvement >1.2 and a present score >3.2
  * Non response = Percentage of patients with either an improvement of ≤0.6 or an improvement >0.6 to ≤1.2 and a present score >5.1
Time to onset of benefit | 32 weeks of treatment
  ACR20, will be also analyzed at every clinic visit to allow an analysis of the time to onset of benefit for achievement of ACR
Change in modified van der Heijde Sharp score | 32 weeks of treatment
  • The Sharp method is a composite X-ray scoring system used to assess structural (joint) disease progression in rheumatoid arthritis. The method evaluates both joint erosions (JE) and joint space narrowing (JSN) in bilateral hand and foot joints
Physical function | 32 weeks of treatment
  • Improvement in physical function is assessed by change from baseline in HAQ (Health Assessment Questionnaire) at Week 32.The HAQ-DI (disability index) is composed of 8 categories as follows: dressing and grooming, arising, eating, walking, hygiene, reach, grip and activities, for which there are at least 2 questions by category. The patient will be asked to score how difficult he/she feels it is to perform such activities using a 0 to 3 scoring (0=without any difficulty, 1=with some difficulty, 2=with much difficulty and 3=unable to do). If the patient is using assistance for any of these activities, scoring may be adjusted. For each category, the highest score given for one of the question is attributed to the category. The total score is the sum of all categories' scores divided by the number of answered categories (at least 3 categories should be answered)
Functional Assessment of Chronic Illness Therapy Fatigue scale (FACIT-Fatigue) | 32 weeks of treatment
  The FACIT-Fatigue is a 13-item questionnaire rated 0 to 4. The patient will be asked to answer to 13 questions rated 0 to 4 (0=not at all,
  1=a little bit, 2=some what, 3=quite a bit, 4=very much
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]). | 32 weeks of treatment
  Infections, hematological disorders, neurologic disorders and malignancies. Adverse Drug Reactions. Incidence, seriousness and severity. Serum Hematological and chemistry values.Local Adverse Drug Reactions
Steady state concentration | At week 16 and 32
  Etanercept concentration measure
Immunogenicity | At week 16 and 32
  Antibodies anti-Etanercept measure

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Velasco, MD, Principal Investigator — Instituto Médico CER; Maria de los Angeles Correa, MD, Principal Investigator — PAMPA; Maria Alicia Lazaro, MD, Principal Investigator — IARI; Rodolfo Pardo Hidalgo, MD, Principal Investigator — CER San Juan; Daniel Siri, MD, Principal Investigator — CAICI; Alberto Jorge Spindler, MD, Principal Investigator — Centro Médico Privado de Reumatología; Ingrid Strusberg, MD, Principal Investigator — Centro Reumatologico Strusberg; Patricio Tate, MD, Principal Investigator — OMI; Horacio Oscar Venarotti, MD, Principal Investigator — Atención Integral en Reumatología
Locations (1):
- Instituto Medico CER, Bs As, Argentina

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Strusberg I, Mysler E, Citera G, Siri D, de Los Angeles Correa M, Lazaro MA, Pardo Hidalgo R, Spindler A, Tate P, Venarotti H, Velasco Zamora J, Klimovsky E, Federico A, Scheines E, Gonzalez E, Cordeiro L, Lago N. Efficacy, Safety, and Immunogenicity of Biosimilar Etanercept (Enerceptan) Versus Its Original Form in Combination With Methotrexate in Patients With Rheumatoid Arthritis: A Randomized, Multicenter, Evaluator-Blinded, Noninferiority Study. J Clin Rheumatol. 2021 Sep 1;27(6S):S173-S179. doi: 10.1097/RHU.0000000000001616. PMID 33337815